CLINICAL TRIAL: NCT01103232
Title: Cross-Education Of Muscular Strength: Is Cross-Training Effects Confined To Untrained Contralateral Homologous Muscle
Brief Title: Cross-Education Of Contralateral Antagonists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vakif Gureba Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ILHAN KARACAN, Chief of Physical Med & Rehab Clinic, Vakif Gureba Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: VGEAH FTR
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Muscle Strength Quantitative Trait Locus 1
Keywords: Cross education; Muscle training
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrical Muscle Stimulation (Experimental): Electrical muscle stimulation of the right wrist flexor muscles was applied
  Interventions: Procedure: Experimental group
- Control (Sham Comparator): Transcutaneous electrical nerve stimulation was applied
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Experimental group — Electrical muscle stimulation (EMS) of the right wrist flexor muscles was applied. EMS was applied for 20 minutes. Maximum current intensity tolerated was used so as to stimulate the highest possible number of motor unit. The stimulation intensity increased every five minutes during a session. Electrical stimulation was applied for thirty sessions (one session a day, five days a week for six weeks.)
  Other Names: Electrical Muscle Stimulation
  Arms: Electrical Muscle Stimulation
Procedure: Control group — Conventional mode of transcutaneous electrical nerve stimulation (TENS) was applied for the control subjects. TENS was applied for 20 minutes. The stimulus intensity was adjusted as the lowest current at which the subject felt only a slight tickling of the impulses. A visible, and palpable muscle contraction was not provided during TENS stimulation. The stimulus intensity was not changed during the first session. Subsequently, TENS was applied at same intensity in all sessions. TENS was applied for thirty sessions (one session a day, five days a week for six weeks).
  Other Names: Transcutaneous electrical muscle stimulation
  Arms: Control

SUMMARY:
Previous studies well documented the impact of unilateral training of limb muscle on the untrained contralateral homologous muscle. The aim of this study is to evaluate whether the electrical muscle stimulation on the dominant wrist flexors for 6 weeks cause an increase in the muscle strength of the contralateral wrist extensors in healthy adult men.

Ethical approval was obtained from Institutional Review Board. All participants were volunteers and provided written informed consent. Among young adult males working in our hospital, 30 subjects who voluntarily accepted to participate in this study were assessed for eligibility. Twenty three young-adult healthy males were included in this double-blind prospective study. These volunteers were randomized into two groups. In Electrical Muscle Stimulation (EMS) group, electrical muscle stimulation of the right wrist flexor muscles was applied; in Controls, transcutaneous electrical nerve stimulation was applied. Electrodes were placed over the flexor aspect of the right forearm in both groups. Electrical stimulation was applied for thirty sessions (one session a day, five days a week for six weeks) in both groups by the same researcher. Compex2 (Medicompex SA, Switzerland) was used for electrical stimulation. Isokinetic torque was measured in the right and left wrist flexors and extensors before and after trial. Isokinetic torque was measured in the right (trained) and left (untrained) forearm with the Cybex (Humac 2004/Norm) extremity-testing system.

DETAILED DESCRIPTION:
It has been reported that strength training of unilateral limb causes an increase in voluntary strength not only in the trained limb, but also in the contralateral untrained limb. This phenomenon is known as "cross-education, cross-training or contralateral strength training effect" . Cross-education of muscle strength can occur in both upper and lower limb muscles.It is not gender and age specific and can occur with training accomplished by voluntary effort, electrical stimulation of muscles or mental practice of unilateral contractions. Electrostimulation is one of the most efficient methods to induce cross-education.

Although it is clear that unilateral training has a contralateral effect, the mechanisms behind this effect remain unclear. Because of the specific nature of cross education, modification in neural function is the more likely mechanism underlying this effect. The potential neural mechanisms can be broadly categorized as either ''central" or ''peripheral (spinal)" adaptations. Central neural mechanisms involved in the excitation of the relevant part of the cortex during voluntary contraction of the trained limb are thought to produce contralateral facilitation. The cross-extension reflex is the primary spinal neural mechanism for cross-education.

In the studies performed up today, the contralateral effects of unilateral training were evaluated in the contralateral homologous muscles. However it's not reported whether a change in the muscle strength have been observed in the antagonists of the contralateral homologous muscles. In a study, after one session of unilateral surface electrical stimulation of the rectus femoris, an increase in the isometric force and EMG activity of the contralateral rectus femoris, but a decrease in the EMG activity of the contralateral biceps femoris was reported in adult men. It's proposed that, the EMG activity decrease in the biceps femoris may be explained by cross-extension reflex. The effect of long-time exercise or electrical muscle stimulation on the antagonists of the contralateral homologous muscles is not clear.

The aim of this study is to evaluate whether the electrical muscle stimulation on the dominant wrist flexors for 6 weeks cause an increase in the muscle strength of the contralateral wrist extensors in healthy adult men.

ELIGIBILITY:
Inclusion Criteria:

* young-adult healthy volunteer
* male
* right hand dominant

Exclusion Criteria:

* a chronic disease such as metabolic/endocrine bone disease (osteoporosis, osteomalacia, paget's disease etc)
* myopathy
* tendinopathy
* neurologic disorders (hypoesthesia/anesthesia, epilepsy, paralysis)
* dermatologic disease
* peripheral vascular disease
* joint disease
* cardiac pacemaker
* noncooperative
* professional sportsman
* regular sportive activity such as tennis, volleyball
* heavy worker

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ILHAN KARACAN, MD, Study Chair — Vakif Gureba Training & Research Hospital

REFERENCES:
- [Derived] Sariyildiz M, Karacan I, Rezvani A, Ergin O, Cidem M. Cross-education of muscle strength: cross-training effects are not confined to untrained contralateral homologous muscle. Scand J Med Sci Sports. 2011 Dec;21(6):e359-64. doi: 10.1111/j.1600-0838.2011.01311.x. Epub 2011 Apr 18. PMID 21496110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All cases were recruited within 6 weeks in the VGEAH PMR Clinic
Groups:
- Experimental: Electrical muscle stimulation of the right wrist flexor muscles was applied
Period: Overall Study
Arm/Group | Experimental | Control
Started | 13 | 13
Completed | 12 | 11
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.6 (5.7) | 34.2 (4.8) | 32 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 13 | 26
Muscle strength [Mean (Standard Deviation); unit: Newton meters] | 44.1 (12.0) | 11.7 (6.3) | 33.2 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Muscle Strength in the Contralateral Untrained Wrist Muscles
Description: Isokinetic torque was measured in the contralateral untrained wrist muscles with the Cybex (Humac 2004/Norm) extremity-testing system before and after experiment.
Time Frame: 6 weeks (The change calculated as 6 months minus baseline)
Measure: Mean (Standard Deviation); unit: Newton meters
Arm/Group | Experimental | Control
Number analyzed (Participants) | 13 | 13
Newton meters | 44.1 (12.0) | 11.7 (6.3)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: 8 weeks
Arm/Group | Experimental | Control
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
This study has small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No